CLINICAL TRIAL: NCT07304414
Title: Clinical Improvement Following Optokinetic Stimulation in Mal de Débarquement Syndrome: A Case Study
Brief Title: Optokinetic Stimulation in Mal de Debarquement Syndrome: Case Report
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, gorkem ata, PT Ph.D., Istanbul Medipol University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-6657
Record Dates: First submitted 2025-12-08; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Mal de Debarquement Syndrome (MdDS)
Keywords: mal de debarquement syndrome; optokinetic stimulation; dizziness; postural balance; quality of life; vestibular disorders
MeSH Terms: conditions — Mal de debarquement; Dizziness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Optokinetic stimulation (OKS) Intervention (Experimental): The participant will receive optokinetic stimulation. The intervention consists of full-field visual stimulation with horizontally moving stripes synchronized with slow head roll movements at a frequency of 0.167 Hz (10 bpm). Sessions will be performed online via the Smart Optometry application, twice daily for 5 consecutive days, with each session lasting approximately 4 minutes. The goal of the intervention is to recalibrate vestibulo-ocular reflex activity and reduce dizziness and imbalance symptoms associated with Mal de Débarquement Syndrome.
  Interventions: Other: Optokinetic stimulation

INTERVENTIONS:
Other: Optokinetic stimulation — The planned optokinetic stimulation (OKS) application will be implemented. The application will last for 5 consecutive days, with a total of 4 sessions, two in the morning and two in the afternoon. Each session will last 5 minutes, and head turns will be synchronized with a metronome at 10 beats per minute (10 bpm). Each beat will complete a full right-left cycle, achieving a frequency of approximately 0.167 Hz. This arrangement reflects the standardized protocol recommended in the literature.
  The application will be conducted online, and the participant will use the "Optokinetic nystagmus (OKN) lines" section within the "Smart Optometry" application on their computer. The direction of the lines will move in the direction opposite the patient's dominantly affected side. The participant was seated close to the screen, and approximately 85-90% of their visual field covered by the moving stimuli.

SUMMARY:
This single-case study aims to evaluate the clinical effects of optokinetic stimulation (OKS) on dizziness perception and quality of life in a patient diagnosed with Mal de Débarquement Syndrome (MdDS). The intervention follows a standardized protocol in which the patient performs head roll movements synchronized with optokinetic visual stimulation at a frequency of 0.167 Hz (10 bpm). The study is conducted online using a digital application to provide full-field optokinetic stimulation. The patient's baseline motion sickness susceptibility was characterized using the Motion Sickness Susceptibility Questionnaire-Short Form (MSSQ-SF). Primary outcome measures assessed for change from baseline include the Dizziness Handicap Inventory (DHI), Visual Analog Scale (VAS), and the Istanbul MdDS Scale

DETAILED DESCRIPTION:
Mal de Débarquement Syndrome (MdDS) is a rare neuro-otological disorder characterized by a persistent perception of self-motion, typically described as rocking, swaying, or bobbing sensations, following exposure to passive motion such as sea, air, or land travel. The syndrome can significantly impair balance, spatial orientation, and quality of life. Conventional therapeutic approaches are limited, and symptoms may persist for weeks, months, or even years. Recent studies have suggested that maladaptation of the vestibulo-ocular reflex (VOR) and velocity storage mechanisms may play a central role in the pathophysiology of MdDS.

In this single-case study, a 28-year-old female patient with a clinical diagnosis of MdDS will undergo an online OKS-based rehabilitation program. The intervention will be conducted remotely via the Smart Optometry application, using the "OKN Stripes" module to deliver full-field optokinetic visual stimulation. The participant will sit close to the screen, ensuring that the optokinetic stripes occupy approximately 85-90% of the visual field. The researcher will guide each session online, ensuring the synchronization of head roll movements with the visual stimuli using a metronome (10 bpm). The intervention will be implemented for 3-5 consecutive days, with two sessions in the morning and two in the afternoon, each lasting 4 minutes.

Assessment and Follow-up: Clinical outcomes are evaluated at multiple time points to monitor the progression and long-term sustainability of the treatment:

Baseline (T0): Pre-treatment assessment. Post-treatment (T1): Immediately following the 5-day protocol. Short-term Follow-up (T2): 1 month after treatment. Long-term Follow-up (T3): 1 year after treatment to evaluate the durability of neuroplastic changes.

Primary metrics include the Dizziness Handicap Inventory (DHI) for perceived disability, the Visual Analog Scale (VAS) for dizziness intensity, and the Istanbul MdDS Scale for syndrome-specific symptoms. To determine the patient's clinical profile and support differential diagnosis, the Motion Sickness Susceptibility Questionnaire - Short Form (MSSQ-SF) will be administered initially.

This study aims to contribute to the limited clinical evidence on non-invasive, visual-vestibular rehabilitation strategies for MdDS and to explore the feasibility of delivering optokinetic therapy in an online, remote setting.

ELIGIBILITY:
Inclusion Criteria:

* Subjective perception of movement in the "rocking/bobbing/swaying" type, beginning after exposure to passive motion (sea/aircraft/vehicle, etc.),
* lasting ≥1 month,
* Temporary relief of symptoms upon re-exposure to passive motion,
* Findings not better explained by an alternative diagnosis.
* Head and neck health must be at a level that allows head roll movement during optokinetic stimulation (no serious cervical limitation).

Exclusion Criteria:

* Alternative vestibular/otologic diagnoses: active BPPV, Meniere's disease, acute vestibular neuronitis, significant peripheral vestibulopathy; or significant central cause (stroke, CNS lesion, etc.).
* History of photosensitizer epilepsy or uncontrolled epilepsy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2025-10-24 (Actual); Primary Completion 2025-10-29 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Level of Disability | From enrollment (baseline) until the final follow-up, assessed at multiple time points: baseline, immediately post-treatment (day 5), 1 month, and 1 year.
  Dizziness Handicap Inventory: Provides information about disability and quality of life in individuals with vestibular disorders. The scale assesses the functional, physical, and emotional effects of dizziness on disability over the past month. It consists of 25 questions, 9 functional, 7 physical, and 9 emotional, with three answer options: yes (4 points), sometimes (2 points), and no (0 points). A total score is calculated along with the scores for each subsection. The total score ranges from 0 to 100, with higher scores indicating greater disability. According to the total score, the level of disability is classified as follows: 16-34 points as mild; 36-52 points as moderate; and 54 and above as severe. This scale, whose
Istanbul Mal de Debarquement Scale | From enrollment (baseline) until the final follow-up, assessed at multiple time points: baseline, immediately post-treatment (day 5), 1 month, and 1 year.
  The scale is composed of subfactors to better assess MdDS. The scale consists of four subfactors: "Diagnostic Criteria" (items 1-5), "Dizziness Character" (items 6-9), "Visual Movement Intolerance" (items 10-12), and "Quality of Life" (items 13-18). The scale was designed using a 5-point Likert-type scale, using the terms "Always," "Frequently," "Sometimes," "Rarely," and "Never." These statements were scored from 5 to 1, respectively. The total scale score was calculated as 100. Permission was obtained from the scale's author for use.
Dizziness Severity | From enrollment (baseline) until the final follow-up, assessed at multiple time points: baseline, immediately post-treatment (day 5), 1 month, and 1 year.
  Visual Analog Scale: The participant's dizziness intensity was assessed on a scale between 0 and 10-cm line, where 0 represents "no vertigo/dizziness," and 10 represents "extreme dizziness. Scores are categorized as mild (2-3), moderate (4-5), severe (6-7), quite severe (8-9), and extreme.

CONTACTS AND LOCATIONS:
Overall Officials: Görkem ATA, Ph.D., Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this is a single-patient case study. Sharing de-identified data could risk patient confidentiality. Summary-level data may be reported in future publications.